CLINICAL TRIAL: NCT04060043
Title: Pilot Study to Evaluate the Effects of a New Depot Formulation of Goserelin Acetate 10.8 mg, on Testosterone Levels in Ambulatory Patients With Carcinoma of the Prostate
Brief Title: Pilot Study to Evaluate the Effects of a Generic Goserelin Acetate in Patients With Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CMX Research (Other)
Collaborators: Peptigroupe Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pepti Pro K02
Record Dates: First submitted 2018-07-19; First posted 2019-08-16 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: goserelin; testosterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Goserelin acetate Injection (Experimental): Pepti 10.8mg is a generic formulation of Zoladex® 10.8mg, with the same ingredients (active and excipients), the same formulation, the same dosage, the same size and route of administration.
  Interventions: Drug: Goserelin Acetate

INTERVENTIONS:
Drug: Goserelin Acetate — The Pepti 10.8mg (goserelin acetate) implant is supplied as a cylindrical rod of biodegradable and biocompatible D, L Lactic and glycolic acids copolymer. Each implant contains goserelin acetate equivalent to 10.8mg of goserelin as well as a blend of high and low molecular weight range of D, L lactic and glycolic acids copolymer to total a weight of approximately 36.0mg per depot. The implant will be injected subcutaneously through the patient's anterior abdominal wall.
  Other Names: Pepti 10.8mg; Goserelin acetate implant

SUMMARY:
This open-label study is designed to obtain preliminary data on the efficacy of a new depot formulation of goserelin, Pepti 10.8mg, in ambulatory patients with carcinoma of the prostate who, in the opinion of the Investigator, is a candidate for androgen deprivation therapy, after a single injection. Secondarily, it is designed to assess the pharmacokinetics, safety profile and PSA response of this new formulation.

DETAILED DESCRIPTION:
A 12 week (84 day) single injection study in 12 patients with carcinoma of the prostate.

During the screening phase, all patients will come to the clinic for a screening visit (V1), during which the patient's eligibility will be evaluated and baseline assessments will be performed. Eligible patients will sign the informed consent form at this visit.

Within 2 weeks after the screening visit, eligible patients will receive a subcutaneous injection of Pepti 10.8mg on day 0 (V2) and samples will be collected for goserelin 1h, 1.5h, 2h and 3h after the injection. Monitoring of the effects for approximate 4h after the injection will be performed.

Thereafter, patients will return to the clinic for follow-up visits approximately every 2 weeks (Visit 3 to 9: Day 7, 21, 35, 49, 63, 77 and 84). The follow-up visits are planned to enable repeated blood sampling designed to evaluate the testosterone response, safety profile and PSA response.

ELIGIBILITY:
Inclusion Criteria:

* Be male at least 18 years of age
* Be an ambulatory patient with carcinoma of the prostate (high risk localized or metastatic) documented by available prostate biopsy information, who in the opinion of the treating physician, is a candidate for androgen deprivation therapy
* Have a testosterone level > 1.5ng/mL or >5nmol/L at screening
* Have a life expectancy of at least 1 year
* Have the ability to understand the requirements of the study and is willing to provide written informed consent
* Agree to abide by the study restrictions and return for the required assessments
* only patients who can be discontinued safety from contra-indicated medications discussed in section 7.4 of the protocol can be included in the study

Exclusion Criteria:

* Have brain metastases
* Have vertebral metastases with evidence of spinal cord compression
* Have renal impairment due to ureteric obstruction or a history of obstructive uropathy
* Have excruciating, sever bone pain due to extensive bone metastases (however, concomitant therapy with either flutamide or bicalutamide is permitted and encouraged during the first month of the study, in the case where mile bone metastasis are present or suspected)
* Undergone orchiectomy, adrenalectomy or hypophysectomy
* Have undergone prostatic surgical procedures (e.g. radical prostatectomy, transurethral resection of the prostate) within the last month
* Have undergone localized external beam radiotherapy, brachytherapy, thermotherapy or cryotherapy within the last 4 weeks
* Undergone systemic chemotherapy, immunotherapy (e.g. antibody therapies, tumor-vaccines) or biological response modifiers (e.g. cytokines) within the last 3 months
* Have been treated with 5-alpha-reductase inhibitors (e.g finasteride (Proscar®, Propecia®), dutasteride (Avodart®)) within the last month
* Have been previously treated with luteinizing hormone releasing hormone agonists (LHRHa) (e.g. leuprolide (Lupron®), goserelin (Zoladex®) etc.) except if their testosterone levels are above 5 nmol/L and the patient in a known responder
* Have and ongoing treatment with androgen receptor (AR) blockers (e.g. megestrol (Megace®) or cyproterone (Androcur®). Note: Treatment with bicalutamide (Casodex®) IS permitted.
* Have a known hypersensitivity to gonadotropin releasing hormone (GnRH), GnRH agonists, any Luteinizing Hormone-Releasing Hormone (LHRH) agonists (e.g. leuprolide (Lupron®), goserelin (Zoladex®) etc.) or to the poly(lactic-co-glycolic acid (PLGA)) polymers contained in the study formulation
* Have a liver disease (e.g. cirrhosis, chronic active hepatitis or chronic persistent hepatitis) or has persistent alanine amino-transferase (ALT), aspartate amino-transferase (AST) > 2 X upper limit normal (ULN), serum creatinine > 2 X ULN, serum bilirubin > 2 X ULN
* Have received an investigational drug or participated in a clinical trial within the last 30 days
* Have a clinically serious and/or unstable intercurrent infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy
* Have a body mass index (BMI) < 18.5
* Be an anticoagulated patient with an International Normalized Ratio (INR) ≥ 2
* Have a history of QT prolongation, congenital long QT syndrome, electrolyte abnormalities, Congestive Heart Failure (CHF), or concurrent administration with QT prolonging drugs or QTc > 450 msec

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Changes in testosterone levels | 84 days
  To evaluate the effects of one Pepti implant on testosterone serum concentration from day 0 to day 84

SECONDARY OUTCOMES:
Changes in PSA | 84 days
  To assess the changes in blood PSA (Prostate Specific Antigen) levels from PSA laboratory results. This testing is to be performed to assess whether patients can be considered for continuing treatment with an LHRH analogue.
# of treatment emergent adverse events occurring | 84 days
  To assess the safety profile of depot formulation of Pepti 10.8mg from day 0 to day 84, all adverse events will be recorded.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (5):
  - Exdeo Clinical Research Inc., Abbotsford, British Columbia
  - The Male / Female Health and Research Centre, Barrie, Ontario
  - Jonathan Giddens Medicine Professional Corporation, Brampton, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario
  - Stanley Flax Medical Professional Corporation, Toronto, Ontario
- Georgia (2):
  - Fridon Todua Research Institute of Clinical Medicine, Tbilisi
  - MediClubGeorgia, Tbilisi